CLINICAL TRIAL: NCT02156388
Title: A Single-center, Uncontrolled, Open, Phase 1 Study of Recombinant(Expressed by Pichia Pastoris) Human Serum Albumin/Human Granulocyte-Colony Stimulating Factor(I)Fusion Protein For Injection(GW003)to Metastatic Tumors
Brief Title: Safety and Pharmacokinetic(PK) Study of GW003 to Metastatic Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu T-Mab Biopharma Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Tmab-GW003-NP-01
Record Dates: First submitted 2014-05-28; First posted 2014-06-05 (Estimated); Last update posted 2016-02-24 (Estimated); Status verified 2016-02

CONDITIONS: Chemotherapy-induced Neutropenia; Metastatic Tumors
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (8):
- Ia-GW003 50μg/kg (Experimental): 2-3 subjects
  Interventions: Biological: GW003
- Ia-GW003 150μg/kg (Experimental): 2-3 subjects
  Interventions: Biological: GW003
- Ia-GW003 300μg/kg (Experimental): 3-6 subjects
  Interventions: Biological: GW003
- Ia-GW003 400μg/kg (Experimental): 3-6 subjects
  Interventions: Biological: GW003
- Ia-GW003 500μg/kg (Experimental): 3-6 subjects
  Interventions: Biological: GW003
- Ia-GW003 600μg/kg (Experimental): 3-6 subjects
  Interventions: Biological: GW003
- Ib-GW003 150μg/kg (Experimental): 6-8 subjects
  Interventions: Biological: GW003
- Ib-GW003 300μg/kg (Experimental): 6-8 subjects
  Interventions: Biological: GW003

INTERVENTIONS:
Biological: GW003 — freeze-dried powder；single SC injection

SUMMARY:
This study is designed to access the safety, tolerance and Pharmacokinetic/Pharmacodynamic(PK/PD) of single subcutaneous(SC) injection of GW003 in patients with metastatic tumors.

DETAILED DESCRIPTION:
So far, granulocyte colony stimulating factor (G-CSF) is still currently the only effective and security therapy drug for neutropenia caused by cancer chemotherapy. At present, the widely used G-CSF products are of such short-acting G-CSF product in China. However, there existed some shortcoming about short-acting G-CSF, such as shorter half-life, continuous monitoring of the patient's blood neutrophil count and so on.

Nowadays,long-acting G-CSF product,such as Neulasta®, has become the mainstream of the foreign G-CSF market for its superiority of long half-life and absence of monitoring of the patient's blood neutrophil count. The new drug Recombinant(Expressed by Pichia pastoris) Human Serum Albumin/Human Granulocyte-Colony Stimulating Factor(I)Fusion Protein(GW003) is a long-acting G-CSF.Preclinical studies have shown that GW003 has accelerated neutrophil recovery and can shorten the duration of neutropenia symptoms, also reduce its extent, therefore minimize the likelihood of serious infections, reflecting a better efficacy and more long half-life.

Phase I was performed as two parts, Ia and Ib. Ia was a sequential dose escalation to observe the dose-limiting toxicity(DLT) and Maximum Tolerated Dose of GW003 given subcutaneously to patients without receiving chemotherapy,6 dose cohorts(50、150、300、400、500 and 600μg/kg) with 2-3 subjects in the 50、150μg/kg cohorts and 3-6 subjects（depend on the Dose-limiting toxicity） in the 300、400、500 and 600μg/kg cohorts, to evaluate safety and pharmacokinetics prior to the Ⅰb.

Ib proposed two arms (150 and 300μg/kg；n=6-8/arm), and to determine whether to continue to increase other dose arm based on the safety and efficacy assessment. Subjects need to receive two cycles treatment of AT chemotherapy. In cycle 1, subjects received AT chemotherapy only; in cycle 2, subjects were administered subcutaneously GW003 24 hours after chemotherapy drugs.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with pathologically and/or cytologically-confirmed malignant tumor (phase Ia)
2. Breast-cancer or NSCLC patients are suitable for chemotherapy regimen of receiving docetaxel plus adriamycin and could finish two-cycles adjuvant chemotherapy on schedule
3. 18 years to 65years
4. Patients with Eastern Cooperative Oncology Group(ECOG) performance status 0 or 1 and living at least 6 months
5. No main organ dysfunction, adequate cardiac,hepatic,renal and bone marrow function
6. Adequate hematologic function (value in center laboratory as the standard); white blood cell count (WBC)≥4.0×109/L neutrophil count (ANC)≥1.5×109/L; platelet count (PLT)≥100×109/L; hemoglobin (HGB)≥lOO g/L.
7. Adequate hepatic and renal function(value in center laboratory as the standard):
8. Women of childbearing age need to pregnancy test Prior to receive therapy and agree to use effective contraception throughout the study
9. Subjects, who are willing to follow the study protocol and provide written informed consent voluntarily, have understood the purpose and procedures and could follow requirements of the study

Exclusion Criteria:

1. History of cardiopathy or with signs and symptoms
2. History of bone marrow transplant and/or stem cell transplant
3. Patients with acute infection, systemic anti-infection treatment within 72 hours of study
4. Prior participated in drug therapy, radiotherapy or surgery and other clinical trials within 4 weeks
5. Prior use of recombinant human G-CSF(rhG-CSF)、PEG-rhG-CSF or erythropoietin within 4 weeks of study
6. Patients with history of primary myeloid malignancy or myelodysplasia
7. Known hypersensitivity to test drugs, rhG-CSF or any other biologicals
8. Pregnant female or nursing mother
9. Known HIV positive or active hepatitis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2013-08; Primary Completion 2015-02 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse event | Ia:up to 4weeks;Ib: up to 10weeks
  To evaluate the safety and tolerance of single SC injection of GW003 to Metastatic Tumors.

SECONDARY OUTCOMES:
Duration of severe neutropenia(DSN) | Ia: up to 3weeks;Ib: up to 6weeks.
Anti-GW003 antibody | Ia: up to 28weeks;Ib: up to 34weeks.
  Ia:anti-GW003 antibody was detected pre-dose and when visit,if there exist positive anti-GW003 antibody, another detected should be conducted 6 months after the trial.
  Ib:anti-GW003 antibody was detected pre-dose ,after cycle 2 chemotherapy and when visit,if there exist positive anti-GW003 antibody, another detected should be conducted 6 months after the trial.
half-life(consists of distribution half-life [t1/2α] and elimination half-life [t1/2β]) | Pre-dose、0.5h、1h、2h、3h、6h、9h、12h、24h、48h、72h、96h、120h、144h and 168h post-dose
area under the concentration-time curve (AUC) | Pre-dose、0.5h、1h、2h、3h、6h、9h、12h、24h、48h、72h、96h、120h、144h and 168h post-dose

CONTACTS AND LOCATIONS:
Overall Officials: zhongsheng Tong, Principal Investigator — Tianjin Medical University Cancer Institute and Hospital
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality, China